CLINICAL TRIAL: NCT00904826
Title: An Open Label Study of the Effects of Eculizumab in Neuromyelitis Optica
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sean J. Pittock, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-001240
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2013-11-04 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-08

CONDITIONS: Neuromyelitis Optica; Devic's Disease
Keywords: NMO; Devic's disease; Neuromyelitis optica; NMO-IgG; Aquaporin-4 antibody; Eculizumab; Complement
MeSH Terms: conditions — Neuromyelitis Optica | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eculizumab (Experimental): The patient will receive eculizumab at a dose of 600mg intravenously (an infusion given into the vein) each week for 4 weeks, then 900mg intravenously at the fifth week, then 900mg every 2 weeks for 48 weeks. Subjects will receive therapy for a total of 12 months.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — The patient will receive eculizumab at a dose of 600mg intravenously (an infusion given into the vein) each week for 4 weeks, then 900mg intravenously at the fifth week, then 900mg every 2 weeks for 48 weeks.
  The first infusion will be given at Mayo Clinic site; subsequent infusions will be administered in the subject's home by a company which will send a nurse to administer the infusion. Subjects will receive therapy for a total of 12 months.
  Other Names: Soliris

SUMMARY:
The purpose of this study is to determine if the drug eculizumab reduces the attack rate and improves outcome in patients with neuromyelitis optica.

DETAILED DESCRIPTION:
It has been shown in some scientific studies that the the antibody marker specific for neuromyelitis optica (NMO), known as NMO-Immunoglobulin G (IgG), causes inflammation in brain tissues by activating a substance called complement. Complement can greatly increase the immune attack in the optic nerves (causing optic neuritis (ON)), spinal cords (causing transverse myelitis (TM)) and brains of patients with NMO. Eculizumab has already been shown to be effective in a rare blood disorder known as paroxysmal nocturnal hemoglobinuria (PNH). Attacks of PNH are also mediated through complement. Therefore, the investigators of this study are investigating whether by 'turning off' complement in NMO, further attacks of NMO can be prevented.

The primary (most important) objectives of this study are to determine:

Whether Eculizumab reduces relapse frequency in patients with relapsing NMO. The number of attacks during the one year treatment period will be compared to the number of attacks that occurred prior to initiation of eculizumab treatment. For patients with more than 2 year disease duration, the average number of attacks in the preceding 2 years will be calculated. For patients with less than 2 years disease duration the number of attacks in the preceding year will be used.

The safety profile of eculizumab in patients with NMO.

The secondary objectives are to determine:

Whether eculizumab maintains or improves walking, visual function and quality of life as measured by a variety of established disability scales. We will also assess the severity of an individual attack and the degree of recovery.

How the drug behaves in the patient's blood (called pharmacodynamics and pharmacokinetics).

Depending on our preliminary investigations we may evaluate patient cerebrospinal fluid in the laboratory to see how effective eculizumab is at getting into the cerebrospinal fluid from the blood stream, and to see if the drug reverses the biological effects of the NMO-IgG antibody.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of NMO, as defined by 2006 criteria OR NMO seropositive spectrum disorder (Recurrent ON or longitudinally extensive transverse myelitis (LETM)). All patients must be NMO-IgG seropositive.
2. Clinical evidence of at least 2 relapses in last 6 months or 3 relapses in the last 12 months (with at least 1 relapse occurring in the preceding 6 months).
3. Age ≥18 years
4. Corrected visual acuity 20/100 or better in at least one eye. If fails item # 4 then entry allowed but only if last attack was myelitis and only attacks of myelitis are considered as outcome measurement.
5. Ambulatory (with or without walker). If fails item # 5 then entry allowed but only if last attack was ON and only attacks of ON are considered as outcome measurement.
6. Provision of written informed consent (see attached) to participate in the study.
7. N. meningitidis vaccination at least 14 days prior to receiving the first eculizumab infusion. If patient in midst of an acute relapse, then relapse will be treated with standard therapy and vaccination given only after a minimum of 4 weeks post attack onset.

Exclusion Criteria:

Candidates will be excluded from study entry if any of the following criteria are met at the time of randomization:

1. Progressive neurological deterioration unrelated to relapses of ON or myelitis.
2. Pregnant, breastfeeding, or intending to conceive during the course of the study
3. Patients will not participate in any other clinical therapeutic study or will not have participated in any other experimental treatment study within 30 days of screening
4. Patients with a history of splenectomy, because of a potential increased risk of developing meningococcal infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean J. Pittock, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Background] Wingerchuk DM, Lennon VA, Lucchinetti CF, Pittock SJ, Weinshenker BG. The spectrum of neuromyelitis optica. Lancet Neurol. 2007 Sep;6(9):805-15. doi: 10.1016/S1474-4422(07)70216-8. PMID 17706564
- [Background] Lennon VA, Wingerchuk DM, Kryzer TJ, Pittock SJ, Lucchinetti CF, Fujihara K, Nakashima I, Weinshenker BG. A serum autoantibody marker of neuromyelitis optica: distinction from multiple sclerosis. Lancet. 2004 Dec 11-17;364(9451):2106-12. doi: 10.1016/S0140-6736(04)17551-X. PMID 15589308
- [Background] Lennon VA, Kryzer TJ, Pittock SJ, Verkman AS, Hinson SR. IgG marker of optic-spinal multiple sclerosis binds to the aquaporin-4 water channel. J Exp Med. 2005 Aug 15;202(4):473-7. doi: 10.1084/jem.20050304. Epub 2005 Aug 8. PMID 16087714
- [Background] Wingerchuk DM, Lennon VA, Pittock SJ, Lucchinetti CF, Weinshenker BG. Revised diagnostic criteria for neuromyelitis optica. Neurology. 2006 May 23;66(10):1485-9. doi: 10.1212/01.wnl.0000216139.44259.74. PMID 16717206
- [Background] Hinson SR, Pittock SJ, Lucchinetti CF, Roemer SF, Fryer JP, Kryzer TJ, Lennon VA. Pathogenic potential of IgG binding to water channel extracellular domain in neuromyelitis optica. Neurology. 2007 Dec 11;69(24):2221-31. doi: 10.1212/01.WNL.0000289761.64862.ce. Epub 2007 Oct 10. PMID 17928579
- [Background] Rother RP, Rollins SA, Mojcik CF, Brodsky RA, Bell L. Discovery and development of the complement inhibitor eculizumab for the treatment of paroxysmal nocturnal hemoglobinuria. Nat Biotechnol. 2007 Nov;25(11):1256-64. doi: 10.1038/nbt1344. PMID 17989688
- [Background] Hinson SR, McKeon A, Fryer JP, Apiwattanakul M, Lennon VA, Pittock SJ. Prediction of neuromyelitis optica attack severity by quantitation of complement-mediated injury to aquaporin-4-expressing cells. Arch Neurol. 2009 Sep;66(9):1164-7. doi: 10.1001/archneurol.2009.188. PMID 19752309
- [Result] Pittock SJ, Lennon VA, McKeon A, Mandrekar J, Weinshenker BG, Lucchinetti CF, O'Toole O, Wingerchuk DM. Eculizumab in AQP4-IgG-positive relapsing neuromyelitis optica spectrum disorders: an open-label pilot study. Lancet Neurol. 2013 Jun;12(6):554-62. doi: 10.1016/S1474-4422(13)70076-0. Epub 2013 Apr 26. PMID 23623397

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2009 and November 2010, subjects were directly recruited at the Mayo Clinics in Rochester, Minnesota and Scottsdale, Arizona, or identified through the Mayo Clinic study-specific repository or clinicoserological database.
Period: Overall Study
Arm/Group | Eculizumab
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
Age Continuous [Mean (Full Range); unit: years] | 41.1 [18.4 to 67.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Ethnic origin [Number; unit: participants]
  African American | 2
  Hispanic | 3
  White | 9
Diagnosis [Number; unit: participants]
  Neuromyelitis optica | 8
  Relapsing optic neuritis | 2
  Relapsing transverse myelitis | 4
Coexisting autoimmune diseases [Number; unit: participants]
  Myasthenia gravis | 2
  Idiopathic thrombocytopenic purpura | 2
  Mixed connective tissue disease | 2
  No coexisting autoimmune disease | 10
Type of previous attacks at enrollment [Number; unit: attacks]
  Optic neuritis | 28
  Transverse myelitis | 52
  Brainstem | 1
  Multifocal optic neuritis and transverse myelitis | 3
  Other multifocal | 2
Number of previous attacks per subject [Mean (Full Range); unit: attacks per subject] | 5.5 [2.0 to 10.0]
Expanded Disability Status Scale (EDSS) Score [Mean (Full Range); unit: units on a scale] — The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death) in half-point increments.
  units on a scale | 4.8 [2.0 to 8.0]

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Neuromyelitis Optica (NMO) Attacks Per Year
Time Frame: baseline, after 12 months of treatment
Measure: Median (Full Range); unit: attacks per year
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
attacks per year
  Baseline | 3 [2 to 4]
  After 12 months of treatment | 0 [0 to 1]
Statistical Analysis 1: Comparison: Eculizumab; Comparison between before treatment and one year after treatment; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number Subjects Experiencing an NMO Attack in 12 Months of Eculizumab Treatment
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
participants | 2

3. Secondary Outcome: Change in Expanded Disability Status Scale (EDDS) Score
Description: The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death) in half-point increments.
Time Frame: baseline, 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
units on a scale | -0.7 [-1.2 to -0.2]
Statistical Analysis 1: Comparison: Eculizumab; Comparison was made between baseline and after 12 months of treatment; Test type: Superiority or Other; p = 0.0078, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Subjects With Change in Visual Acuity in at Least One Eye by at Least One Point
Description: Visual acuity was measured using the the Visual Acuity subscale of the Opticospinal Impairment Score (OSIS) for Exacerbations. This subscale ranges from 0 (normal) to 8 (no light perception).
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
participants | 5

5. Secondary Outcome: Number of Subjects With Change in Ambulation by at Least 1 Point
Description: Ambulation was measured by the Hauser Ambulation Index, which ranges from 0 (asymptomatic; fully active) to 9 (restricted to wheelchair; unable to transfer self independently.)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
participants | 3

6. Secondary Outcome: Mean Serum Concentration of Eculizumab
Time Frame: 6 weeks, 3 months, 6 months, 9 months, 12 months
Population: Patient 13 was excluded from the 3 months measurement because she had temporarily discontinued treatment.
Measure: Mean (Standard Deviation); unit: micrograms/mL
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
micrograms/mL
  6 weeks | 206 (77)
  3 months | 187 (91.2)
  9 months | 230 (85.3)
  12 months | 246 (102)

7. Secondary Outcome: Percentage Hemolysis
Description: Percentage of hemolysis is a measure of complement activity. Less than 20% lysis is deemed to be complete complement inhibition.
Time Frame: baseline, 6 weeks, 3 months, 6 months, 9 months, 12 months
Population: Subject 13 was excluded at 3 months visit because she had temporarily discontinued treatment.
Measure: Mean (Standard Deviation); unit: percentage of hemolysis
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
percentage of hemolysis
  Baseline | 88.5 (13.2)
  6 weeks | 0.4 (0.8)
  3 months | 0 (0)
  6 months | 0.2 (0.6)
  9 months | 0.4 (0.9)
  12 months | 0.9 (1.5)
Statistical Analysis 1: Comparison: Eculizumab; Comparison is between 6 weeks and baseline; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Eculizumab; Comparison is between 3 months and baseline; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Eculizumab; Comparison is between 6 months and baseline; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Eculizumab; Comparison is between 9 months and baseline; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Eculizumab; Comparison is between 12 months and baseline; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Mean Eculizumab Concentration in Cerebrospinal Fluid (CSF)
Time Frame: 3 months
Population: 12 subjects including subject 13 agreed to have CSF draw at the 3 month visit, but subject 13 was excluded because she had temporarily discontinued treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eculizumab
Number analyzed (Participants) | 11
ng/mL | 34.7 (18.7)

9. Secondary Outcome: Mean Complement Protein 5 (C5) Concentration in CSF
Time Frame: baseline, 3 months
Population: At 3 months, C5 was undetectable in 6 subjects; patient 13 was excluded because she had temporarily discontinued treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eculizumab
Number analyzed (Participants) | 14
ng/mL
  Baseline | 144 (75.5)
  3 months | 60.8 (23.3)
Statistical Analysis 1: Comparison: Eculizumab; Comparison was between 3 months and baseline; Test type: Superiority or Other; p = 0.0019, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Eculizumab
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=14)
Meningococcal infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=14)
Headache (General disorders) | 9 (23)
Nausea (Gastrointestinal disorders) | 6 (18)
Dizziness (General disorders) | 6 (13)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Coughing (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Abdominal Pain (General disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (9)
Urinary tract infection (Infections and infestations) | 2 (6)
Flu like symptoms (General disorders) | 2 (3)
Swelling or ankle swelling (Blood and lymphatic system disorders) | 2 (2)
Fatigue (General disorders) | 2 (3)
Nasal congestion or watery eyes (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No